CLINICAL TRIAL: NCT00701818
Title: Coronary Arteriosclerosis in Patients With Acute Ischemic Stroke Prevalence and Characteristics as Measured by CT Angiography, Echocardiography and Biomarkers
Brief Title: Coronary Arteriosclerosis in Patients With Acute Ischemic Stroke
Acronym: CORAIS
Status: Completed | Type: Observational
Sponsor: Vejle Hospital (Other)
Responsible Party: Principal Investigator, Jesper K. Jensen, Md, Vejle Hospital
Other Study IDs: S-20070097
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Ischemic Stroke; Myocardial Ischemia; Coronary Arteriosclerosis
MeSH Terms: conditions — Ischemic Stroke; Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The specific objectives of this thesis are in a cohort of patients with an acute ischemic stroke,

1. To establish the degree of coronary arteriosclerosis.
2. To describe left ventricular systolic and diastolic function in relation to changes of NT-proBNP.

DETAILED DESCRIPTION:
Background:

Stroke and myocardial infarction are leading causes of death and disability in the industrialized countries. Multiple interactions exist between the various forms of cardiovascular and cerebrovascular diseases and several risk factors for the development of stroke and major cardiovascular diseases are similar, as emphasized by the recent publication of a common set of guidelines for the primary prevention of both. Following myocardial infarction the stroke incidence is markedly increased, particular early after myocardial infarction. Additionally, non-stroke cardiovascular disease, especially coronary artery disease, is the main cause of long-term mortality in patients surviving cerebrovascular diseases. The history of ischemic heart disease in stroke patients is often unreliable because of cognitive and language impairments or simply because ischemic heart disease is asymptomatic. For at least 25 years myocardial damage has repeatedly been proposed as a consequence of an acute stroke, i.e. being neuromediated. Most prior studies were performed in patients with subarachnoid hemorrhage, and consequently only limited data regarding ischemic stroke, the most common cerebrovascular ailment, are available. Recently it has been demonstrated that highly sensitive and specific markers for the detection of myocardial necrosis, i.e., cardiac troponins, may be elevated in 0 % - 34 % of patients with ischemic stroke. However, the majority of the studies conducted have not sufficiently evaluated coexisting coronary artery disease. The neuromediated theory has been supported in patients with subarachnoid hemorrhage and elevated troponin levels due to lack of significant obstructive coronary artery disease evaluated by coronary angiograms. Little is known about a conceivable cause-effect relationship between acute ischemic stroke and myocardial necrosis, i.e., neuromediation, or if the elevated levels of troponin are caused by direct cardiac damage, i.e., AMI.

Recently, several reports have demonstrated that levels of natriuretic peptides are increased in patients with acute ischemic stroke. The hormone Brain Natriuretic Peptide (BNP) and its split product (NT-proBNP) derives predominantly from the myocardium and is processed as a response to stretch of cardiomyocytes and hemodynamic stress. The mechanism of elevated levels of NT-proBNP in the setting of acute ischemic stroke is unknown. Myocardial ischemia is known to cause release of NT-proBNP. Accordingly, levels of NT-proBNP are higher in acute ischemic stroke patients with ST-segment depression on 12-lead ECG than in those without. However, it is unknown whether levels of NT-proBNP are correlated to coronary arteriosclerosis and left ventricle function in patients with acute ischemic stroke.

The current gold standard for the detection of atherosclerotic coronary artery disease (CAD), invasive coronary angiography (CAG), allows direct visualization of the coronary artery lumen. Inconvenience to patients and a small but not negligible risk of complications related to CAG have prompted an intensive search for alternative, reliable non-invasive means of coronary artery visualisation. Standard non-invasive methods such as stress testing lack sufficient sensitivity in detecting significant CAD. Over the last decade multislice computed tomography (MSCT) has emerged as a promising non-invasive method in the assessment of CAD. Previous studies have convincingly demonstrated a very high negative predictive value of MSCT coronary angiography (CTA) with CAG as the reference. Thus, a normal CTA seems to allow the clinician to rule out the presence of hemodynamic relevant coronary artery stenoses with a high degree of reliability. In addition to detecting significant coronary artery stenosis, recent focus has been on visualising and characterising coronary artery plaques. Both necropsy and coronary intravascular ultrasound (IVUS) studies have shown that "normal" vessels at CAG may in fact contain a significant amount of atherosclerotic plaques. Independent of the degree of coronary artery stenosis, some plaques may be at increased risk of erosion or rupture. The latter, unstable plaques are thought to trigger acute coronary ischemic events. Accordingly, the release of troponins, NT-proBNP and ECG changes observed in these patients could be due to CAD. So far serial investigation of CAD has never been performed in patients with acute ischemic stroke.

Objective:

The specific objectives of this thesis are in a cohort of patients with an acute ischemic stroke,

1. To establish the degree of coronary arteriosclerosis.
2. To describe left ventricular systolic and diastolic function in relation to changes of NT-proBNP.

Inclusion Criteria:

1. Age ≥ 18 years old
2. Symptoms suggestive of an acute ischemic stroke
3. Informed consent

Exclusion Criteria:

1. Present intracerebral or subarachnoid haemorrhage
2. Present intracerebral vascular malformation
3. Present transient ischemic attack
4. Prior coronary bypass surgery or percutaneous coronary intervention
5. Pacemaker
6. Allergy to contrast
7. Lack of cooperation

Clinical evaluation:

All patients included in the study will have a computed tomography scan performed at the time of admission. The patients included undergo a baseline clinical evaluation, a structured interview and examination of medical records focusing at

* Hypertension
* Dyslipidemia
* Diabetes mellitus
* Smoking
* Alcohol consumption
* Medication
* Atrial fibrillation
* Ischemic heart disease
* Angina Pectoris (CCS classification)
* Heart failure (NYHA- and KILLIP-classification)
* Peripheral Arterial Occlusive Disease

Electrocardiography:

A 12-lead resting ECG is obtained immediately on admission and up to each of the following five days in the morning. The 12-lead resting ECGs were recorded in the supine position with a paper speed of 25 mm/s. All ECGs are interpreted by two experienced cardiologist under blinded conditions. The ECG findings of interest in this thesis are horizontal or downsloping ST-segment depression ≥0.1 mV, T-wave inversion ≥0.1 mV in two or more contiguous leads, and ST-segment elevation ≥0.2 mV in leads V1-3; ST-elevation ≥0.1 mV in other leads.

Holter monitoring:

Holter 24-hour ECG recordings are performed with Reynolds Medical Tracker 3 and a Pathfinder 700 (Reynolds Medical Limited, England) for analysis. An ischemic episode is defined as ≥0.1 mV of horizontal or downsloping ST-segment depression compared to baseline, measured 80 ms after the J-point. An episode of ST-segment depression has to last ≥2 minutes in order to count and two episodes have to be separated by at least two minutes. In patients with resting ST-segment depression additional ≥0.1 mV ST-segment depression has to be present. Every episode of ST-segment deviation is verified by ECG printouts (25 mm/s). Furthermore, Holter monitoring will be analyzed for occurrence of atrial arrhythmias. Evaluation of ischemic and arrhythmias episodes is interpreted visually by two cardiologist blinded to other patient characteristics.

Blood Sampling:

Blood samples are drawn immediately on admission and up to each of the following five days in the morning. Specimens for NT-proBNP, troponin T and I, CK-MB, myeloperoxidase, oxidated low-density lipoprotein, osteoprotegerin are collected. All analyses are performed at the Department of Clinical Biochemistry, Vejle Hospital.

Echocardiography:

Doppler echocardiography will be performed as soon as the patient condition allows. Examinations will be performed on a GE medical Vivid 7 ultrasound machine. Images will be obtained from the parasternal and apical windows. M-mode recordings will be done in the parasternal long-axis view. Pulsed Doppler measurements of mitral inflow will be obtained with the transducer in the apical four-chamber view, with a 1-2 mm Doppler sample volume placed between the tips of mitral leaflets during diastole. Tissue Doppler imaging of the mitral annulus will be obtained from the apical 4-chamber view with a 1.5-mm sample volume placed at the medial mitral annulus. All Doppler echocardiographic examinations are done with horizontal sweep set to 100 mm/s. At least 3-5 cardiac cycles will be measured. Finally color coded real time tissue Doppler images will be acquired in the apical windows.

* End-systolic, end-diastolic volume and ejection fraction will be calculated according to the Simpson modified biplane method.
* LV mass will be estimated using the recommendations of the American Society of Echocardiography.
* Maximal left atrial volume will be measured at end-systole with the use of two orthogonal apical views.
* From the pulsed wave mitral inflow signal, peak E wave velocity, peak A wave velocity, and mitral E-wave deceleration time will be measured. From pulsed wave Doppler recording of LV outflow ejection time will be recorded. From these recordings Tei index will be assessed.
* From peak tricuspid regurgitant velocity and size of inferior v. cava pulmonary arterial systolic pressure will be estimated.
* From the tissue Doppler assessment of the medial mitral annulus early (E') diastolic velocity will be recorded. Diastolic function will be graded in grades 0-3 and diastolic E/e' ratio calculated.
* From color coded tissue Doppler images systolic longitudinal fibre shortening will be assessed using tissue tracking, and systolic strain will be assessed on a regional basis.

Multislice computed tomography coronary angiography:

Examinations are performed at the Department of Cardiology, Vejle Hospital with dual source CT (DSCT) scanner technology (Siemens Definition; Forcheim, Germany). Tube voltage is 120kV for both tubes, current 560 mA with modulation and full current between 25 % - 80 % of the RR interval. Gantry rotation time is 330 msec, pitch is 0.20-0.44 according to the heart rate. Per rotation 64 slices are generated with a collimation of 0.6 mm resulting in an isotropic voxel size of approximately 0.6 mm. A bodyweight adapted volume of contrast agent (Iomeron 350) is injected continuously at rate of 5 ml /sec. The scan is initiated according to a bolus tracking protocol (aortic root attenuation level of 100 HU). Axial images are reconstructed with 0.75 mm slice thickness, and a 0.5 mm increment using a medium sharp kernel (B26) and retrospective ECG gating. The reconstructions are performed in 5 % steps over the relevant part of the RR cycle using a single-segment algorithm. In case of atrial fibrillation, data sets were reconstructed in 50 ms steps. Using a semi-automated Hounsfield dependent algorithm, differentiation between contrast enhanced lumen, vessel wall and atherosclerotic plaques, is performed. Atherosclerotic plaques will be categorized into calcified (>130 HU, high density plaque), non-calcified (< 60 HU, low density plaque), and mixed-type plaques (60-130 HU, intermediate density plaque), respectively. According to an American Heart Association 17 segmental coronary artery model, stenoses > 50 % or > 75 % are registered. Main coronary vessels (left main, left anterior descending artery, circumflex, and the right coronary artery) and side branches with a lumen diameter > 1, 5 mm are analysed. Image quality will be assessed as good (no artefacts related to motion, calcification or noise), satisfactory (artefacts present, but assessment of artery stenosis possible), or unsatisfactory (artefacts compromising the evaluation of artery stenosis). Images are analysed by two independent observes without knowledge of the patient history.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Symptoms suggestive of an acute ischemic stroke
3. Informed consent

Exclusion Criteria:

1. Present intracerebral or subarachnoid haemorrhage
2. Present intracerebral vascular malformation
3. Present transient ischemic attack
4. Prior coronary bypass surgery or percutaneous coronary intervention
5. Pacemaker
6. Allergy to contrast
7. Lack of cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is a prospective, consecutive study of patients primarily admitted to the Department of Neurology, Vejle Hospital with symptoms suggestive of an acute ischemic stroke according to the World Health Organization criteria
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Steffensen, MD, PhD, Study Chair — Vejle Hospital; Dan Atar, MD, DMSci, Study Chair — Division of Cardiology, Aker University Hospital, University of Oslo, Norway; Jens O Kjærsgaard, MD, Study Chair — Department of Neurology, Vejle Hospital, Denmark; Ivan Brandslund, MD, DMSCi, Study Chair — Department of Clnical Biochemistry, Vejle Hospital, Denmark
Locations (1):
- Department of Cardiology, Vejle Hospital, Vejle, Denmark

REFERENCES:
- [Background] Goldstein DS. The electrocardiogram in stroke: relationship to pathophysiological type and comparison with prior tracings. Stroke. 1979 May-Jun;10(3):253-9. doi: 10.1161/01.str.10.3.253. PMID 462510
- [Background] Lindgren A, Wohlfart B, Pahlm O, Johansson BB. Electrocardiographic changes in stroke patients without primary heart disease. Clin Physiol. 1994 Mar;14(2):223-31. doi: 10.1111/j.1475-097x.1994.tb00508.x. PMID 8205753
- [Background] Dimant J, Grob D. Electrocardiographic changes and myocardial damage in patients with acute cerebrovascular accidents. Stroke. 1977 Jul-Aug;8(4):448-55. doi: 10.1161/01.str.8.4.448. PMID 898240
- [Background] Khechinashvili G, Asplund K. Electrocardiographic changes in patients with acute stroke: a systematic review. Cerebrovasc Dis. 2002;14(2):67-76. doi: 10.1159/000064733. PMID 12187009
- [Background] Barber M, Morton JJ, Macfarlane PW, Barlow N, Roditi G, Stott DJ. Elevated troponin levels are associated with sympathoadrenal activation in acute ischaemic stroke. Cerebrovasc Dis. 2007;23(4):260-6. doi: 10.1159/000098325. Epub 2006 Dec 29. PMID 17199083
- [Background] Jensen JK, Atar D, Mickley H. Mechanism of troponin elevations in patients with acute ischemic stroke. Am J Cardiol. 2007 Mar 15;99(6):867-70. doi: 10.1016/j.amjcard.2006.10.052. Epub 2007 Feb 2. PMID 17350385
- [Background] Jensen JK, Kristensen SR, Bak S, Atar D, Hoilund-Carlsen PF, Mickley H. Frequency and significance of troponin T elevation in acute ischemic stroke. Am J Cardiol. 2007 Jan 1;99(1):108-12. doi: 10.1016/j.amjcard.2006.07.071. Epub 2006 Nov 9. PMID 17196472
- [Background] Fure B, Bruun Wyller T, Thommessen B. Electrocardiographic and troponin T changes in acute ischaemic stroke. J Intern Med. 2006 Jun;259(6):592-7. doi: 10.1111/j.1365-2796.2006.01639.x. PMID 16704560
- [Background] Etgen T, Baum H, Sander K, Sander D. Cardiac troponins and N-terminal pro-brain natriuretic peptide in acute ischemic stroke do not relate to clinical prognosis. Stroke. 2005 Feb;36(2):270-5. doi: 10.1161/01.STR.0000151364.19066.a1. Epub 2004 Dec 16. PMID 15604421
- [Background] Jensen JK, Mickley H, Bak S, Korsholm L, Kristensen SR. Serial measurements of N-terminal pro-brain natriuretic peptide after acute ischemic stroke. Cerebrovasc Dis. 2006;22(5-6):439-44. doi: 10.1159/000094997. Epub 2006 Aug 11. PMID 16912478
- [Background] Iltumur K, Yavavli A, Apak I, Ariturk Z, Toprak N. Elevated plasma N-terminal pro-brain natriuretic peptide levels in acute ischemic stroke. Am Heart J. 2006 May;151(5):1115-22. doi: 10.1016/j.ahj.2005.05.022. PMID 16644347
- [Background] Jensen JK, Korsholm L, Hoilund-Carlsen PF, Atar D, Kristensen SR, Mickley H. The relation between electrocardiographic ST-T changes and NT-proBNP in patients with acute ischemic stroke. Scand Cardiovasc J. 2007 Oct;41(5):294-8. doi: 10.1080/14017430701601644. PMID 17886116